CLINICAL TRIAL: NCT01416259
Title: A Randomized, Placebo-Controlled, Four-Period Crossover Definitive QT Study Of The Effects of APF530 Exposure, High-Dose IV Granisetron and Moxifloxacin on QTc Prolongation
Brief Title: A Phase I Study of the Effects of APF530 Exposure, Granisetron and Moxifloxacin
Status: Completed | Type: Observational
Sponsor: Heron Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: APPA C2011-01
Record Dates: First submitted 2011-08-10; First posted 2011-08-15 (Estimated); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Healthy
Keywords: QTc Prolongation
MeSH Terms: interventions — Withholding Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- APF530 Exposure, Granisetron and Moxifloxacin, Placebo: Arm 1:APF530 Exposure Arm 2:Granisetron IV Arm 3:Moxifloxacin Arm 4:Placebo
  Interventions: Drug: Withdraw treatment

INTERVENTIONS:
Drug: Withdraw treatment

SUMMARY:
This Phase I study will be performed in a double-blind, randomized, crossover design in healthy male and female subjects. The central ECG laboratory will be blinded to treatment. Every effort will be made to enroll equal numbers of males and females into the study.

Eligible subjects will participate in a screening phase (within 28 days of the dosing day), a treatment phase and a final visit, which will be conducted on discharge from the study. Study duration will be 32 days with a total of approximately 12 days of confinement. During the resting ECG periods, 12-lead digital ECGs will be extracted from continuous telemetry at selected time points to assess potential ECG effects. Blood samples for PK evaluation will be collected in conjunction with the ECG time points.

ELIGIBILITY:
Inclusion Criteria:

* Subjects in good health
* aged between 18-50 years
* weigh at least 50 kg (110 pounds)
* have a body mass index of 18-32 kg/m2 inclusive
* capable of understanding and complying with the protocol
* have signed the informed consent

Exclusion Criteria:

* have a history of drug abuse or are current smokers
* have a known hypersensitivity to Moxifloxacin or granisetron
* a history or presence of clinically significant abnormal 12-lead ECG or an ECG with QTc by Bazett's correction of > 450 ms in men, > 470 ms in women on the screening ECG
* PR > 240 ms, QRS > 110 ms or a history of prolongation of QT interval
* a family history of Long QT Syndrome or cardiac disease
* may not have used any medications or consumed any foods contraindicated in the protocol

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Male and Female Subjects
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2011-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
QTc Prolongation | From baseline over 48 hours.
  To evaluate the effect of APF530 given subcutaneously, in normal volunteers, on placebo subtracted change of QTcF

SECONDARY OUTCOMES:
Plasma concentrations of granisetron | From baseline over 48 hours
  To achieve a mean Cmax of granisetron and AUC exposure in normal volunteers equivalent to that achieved by APF530 given subcutaneously, in patients.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Dietz, MD, PhD, Principal Investigator — Spaulding Clinical Research LLC
Locations (1):
- Spaulding Clinical Research, West Bend, Wisconsin, United States